CLINICAL TRIAL: NCT04149015
Title: A Phase II Trial of Neoadjuvant POF in the Treatment of Locally Advanced Gastric Cancer
Brief Title: Neoadjuvant POF in the Treatment of Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNF015
Record Dates: First submitted 2019-10-18; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POF (Experimental): A 3-hour infusion of paclitaxel (135 mg/m2) followed by oxaliplatin (85 mg/m2) and leucovorin (400 mg/m2), administered simultaneously over a 2-hour infusion period. Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating every 14 days for 4 cycles
  Interventions: Drug: paclitaxel ,oxaliplatin,fluorouracil

INTERVENTIONS:
Drug: paclitaxel ,oxaliplatin,fluorouracil — A 3-hour infusion of paclitaxel (135 mg/m2) followed by oxaliplatin (85 mg/m2) and leucovorin (400 mg/m2), administered simultaneously over a 2-hour infusion period. Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating every 14 days for 4 cycles.

SUMMARY:
This study is a single center, phase II study, to evaluate the effectiveness and safety of POF(paclitaxel plus oxaliplatin plus 5-fluorouracil plus leucovorin) , in the neoadjuvant therapy for patients with advanced/metastatic gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old;
* Patients must have histologically or cytologically confirmed resectable gastric or gastroesophageal junction (GEJ) adenocarcinoma without distant metastases. GEJ adenocarcinoma may be classified according to Siewert's classification type I, II, or III
* Patients may have received no prior chemotherapy.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1;
* An expected survival of ≥ 3 months;
* Major organ function has to meet the following criteria; (1) For results of blood routine test:
* Hemoglobin (HB) ≥ 80g / L,
* ANC(absolute neutrophil count) ≥ 1.5 × 109 / L,
* PLT(blood platelet) ≥ 75 × 109 / L, (2) For results of biochemical tests:
* BLT（total bilirubin） ≤ 1.25 times the upper limit of normal (ULN),
* ALT(Alanine aminotransferase) and AST(aspartate aminotransferase ) ≤ 2.5 × ·ULN, liver metastases, if any, the ALT and AST≤ 5 × ULN,
* Serum Cr（creatinine）≤1ULN, Endogenous creatinine clearance rate >50ml/min;
* The patient has a PT（prothrombintime） (INR international normalized ratio) < or = to 1.5 and an PTT（Partial Thromboplastin Time）< than or = to 3 seconds above the upper limits of normal if the patientia t is not on anticoagulation. ·If a patient is on full-dose anticoagulants, the following criteria should be met for enrollment:
* The patient must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin or on stable dose of LMW(Low molecular weight) heparin
* The patient must not have active bleeding or pathological conditions that carry high risk of bleeding (e.g. tumor involving major vessels, known varices)
* Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Ability to understand informed consent and signing of written informed consent document prior to initiation of protocol therapy.

Exclusion Criteria:

1. Subjects with second primary cancer, besides dermatoma, primary cancer of nervous system, non-metastatic prostatic neoplasms.
2. Gastrointestinal bleeding.
3. women of child-bearing age must take a negative result of serum pregnancy test within 7 days prior to enrollment, and willing to use appropriate methods of contraception during the trial and 12 weeks after the last trial drug. For men, who willing to use appropriate methods of contraception during the trial and 12 weeks after the last trial drug.
4. Ongoing corticosteroid drug therapy.
5. With a history of previous severe cardiovascular disease: over grade-two myocardial ischemia or myocardial infarction, congestive hert filure, and myocardial infarction or coagulopathy within 6 months.
6. Having got apoplexy or cardiovascular accident within 6 months.
7. Having got severe peripheral vascular disease in clinics.
8. Subjects who have a history of psychiatric substance abuse and cannot quit or have mental disorders.
9. The researchers concluded that the subjects were not suitable for clinic trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete and subtotal regression (TRG1a/b by Becker) | after 4 cycles (each cycle is 14 days) + surgery; i.e. after 12 weeks in total
  Pathological complete and subtotal regression (TRG1a/b by Becker). TRG1a/b is defined as < 10% residual tumor per tumor bed based on evaluation of the resected esophagogastric specimen in the primary by a pathologist.